CLINICAL TRIAL: NCT01596491
Title: Kind and Duration of Possible Changes of the Sensory Profiles After the Topical Application of Capsaicin (8%) in Patients With Peripheral Neuropathic Pain
Brief Title: Study of Possible Changes in QST After Application of Capsaicin on Patients With Peripheral Neuropathic Pain
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Christoph Maier, Prof. Dr., Head of the Dep. of Pain Management, Ruhr University of Bochum
Other Study IDs: Capsaicin2011
Record Dates: First submitted 2012-02-23; First posted 2012-05-11 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Peripheral Nerve Injury; Postherpetic Neuralgia
Keywords: peripheral nerve injury; postherpetic neuralgia; PNI; PHN; Capsaicin; QST; quantitative sensory testing; sensory profile; neuropathic pain
MeSH Terms: conditions — Peripheral Nerve Injuries; Neuralgia, Postherpetic; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients with peripheral nerve injury: 10 patients with neuropathic pain, because of peripheral nerve injury will obtain a baseline-QST and after capsaicin-application a QST 2, 4, 6, 8 and every 2 weeks until re-occurrence of pain and/or recovery of the capsaicin-induced sensory deficits
  Interventions: Procedure: quantitative sensory testing (QST)
- patients with postherpetic neuralgia: 10 patients with neuropathic pain, because of postherpetic neuralgia will obtain a baseline-QST and after capsaicin-application a QST 2, 4, 6, 8 and every 2 weeks until re-occurrence of pain and/or recovery of the capsaicin-induced sensory deficits
  Interventions: Procedure: quantitative sensory testing (QST)

INTERVENTIONS:
Procedure: quantitative sensory testing (QST) — with QST the small-fibre function is tested by registering thermal and mechanical thresholds, so that changes in the sensory profile can by specified

SUMMARY:
The treatment of neuropathic pain ist still a challenge. A new promising therapy is the use of capsaicin on skin.

The investigators first experiences with capsaicin in patients with peripheral nerve injury showed changes in the sensibility, which achieved its maximal extent after four weeks and was regressive, but not completely abolished 1,5 months after application.

In this study the investigators hope to specify, how long and in which way exactly this changes in sensibility appear.

DETAILED DESCRIPTION:
The topical application of a high dosage of capsaicin (8%) is a new promising approach. There is only little knowledge about the extent and the duration of drug-induced changes of detection and pain thresholds based on a currently recommended standardized quantitative sensory testing (QST). The assessment of QST changes would be an important step forward to understand the way of action as well as the time course of the presumed recovering of the C-fiber function after topical application of a high concentration capsaicin patch.

10 patients suffering from peripheral neuropathic pain due to peripheral nerve injury and 10 patients suffering from postherpetic neuralgia will be investigated by QST following the protocol of DFNS (German Research Network on Neuropathic Pain), using both thermal and mechanical nociceptive as well as non-nociceptive stimuli.

QST will be performed at the following times:

* at baseline
* 2, 4, 6, 8 weeks later, and every two weeks at least until re-occurrence of pain and/or recovering of the capsaicin-induced worsening of the C-fiber function.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years with signed informed consent
* with planned topical application of capsaicin (8%) and with no involvement in any other study
* with neurological proved peripheral neuropathy (e.g. peripheral nerve lesion, postherpetic neuralgia) and with remaining moderate pain intensity under the current treatment (> NRS 3; numeric rating scale 0-10)
* some remaining sensory function at the baseline QST with z-scores ≥ - 3 for cold, warmth and tactile thresholds

Exclusion Criteria:

* with missing informed consent
* with any contraindications for capsaicin application
* with diabetes mellitus,
* using lidocaine patch in the test area in the last 6 months before enrollment
* with inadequate knowledge of the german language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: proved peripheral neuropathy (e.g. peripheral nerve lesion, postherpetic neuralgia)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Duration of the functional loss of the C- and A-delta-fibres after therapeutic application of capsaicin 8% as measured by the impairment of the thermal thresholds | 8 weeks after capsaicin-patch (8%) application
  measurement of thermal detection thresholds for warmth (WDT) and cold (CDT) by QST (standard DFNS protocol), change of z-values for WDT and CDT from baseline to 8 weeks after capsaicin-application (ANOVA)
Extent of the functional loss of the C- and A-delta-fibres after therapeutic application of capsaicin 8% as measured by the impairment of the thermal thresholds | 8 weeks after capsaicin-patch (8%) application
  measurement of thermal detection thresholds for warmth (WDT) and cold (CDT) by QST (standard DFNS protocol), change of z-values for WDT and CDT from baseline to 8 weeks after capsaicin-application (ANOVA)

SECONDARY OUTCOMES:
Decrease of thermal Hyperalgesia | 8 weeks after capsaicin-patch (8%) application
  change of thermal hyperalgesia measured by QST (z-value of heat pain and cold pain threshold)from baseline to 8 weeks after capsaicin-application
Decrease of mechanical hyperalgesia | 8 weeks after capsaicin-patch (8%) application
  change of mechanical hyperalgesia measured by QST (z-value of mechanical pain threshold and mechanical pain sensitivity) from baseline to 8 weeks after capsaicin-application
Decrease of dynamical mechanical allodynia | 8 weeks after capsaicin-patch (8%) application
  change of dynamical mechanical allodynia measured by QST from baseline to 8 weeks after capsaicin-application
Correlation of efficacy on the sensory function and the reported soothing of symptoms after capsaicin-application | 8 weeks after application of capsaicin-patch (8%)
  comparison of z-values for cold, warmth and mechanical detection threshold to the outcome of the german versions of the following questionnaires: PainDETECT, NPSI (Neuropathic Pain Symptom Inventory) and Patient's global impression of change (PGIC), analyzed by ANCOVA

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Maier, Prof.Dr.med, Study Director — University hospital Bergmannsheil department of pain management
Locations (1):
- Bergmannsheil, Department for pain management, Bochum, Germany